CLINICAL TRIAL: NCT01604213
Title: Effects of Vildagliptin/Metformin Combination on Markers of Atherosclerosis, Thrombosis, and Inflammation in Diabetic Patients With Coronary Artery Disease
Brief Title: Effects of Vildagliptin/Metformin Combination on Markers of Atherosclerosis, Thrombosis, and Inflammation in Diabetics With Coronary Artery Disease
Acronym: VAAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Robert Klempfner Heart Rehabilitation Institute, Robert Klempfner MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-12-9455-RK-CTIL
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes Mellitus; Ischemic Heart Disease
Keywords: Type 2 diabetes mellitus; vildagliptin; metformin; atherosclerosis; inflammation; interleukin-6; TNF; atherothrombosis; adiponectin; MMP-9; hs-CRP
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Ischemia; Atherosclerosis; Inflammation; Thrombosis | interventions — Metformin; Vildagliptin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vildagliptin+metformin (Experimental): Oral Vildagliptin+metformin combination
  Interventions: Drug: Metformin plus vildagliptin
- Metformin only (Active Comparator): Oral metformin only
  Interventions: Drug: Metformin only

INTERVENTIONS:
Drug: Metformin plus vildagliptin — Oral Metformin 850mg and vildagliptin 50mg, qd initially, up-titrated to BID if clinically necessary
  Other Names: Eucreas
  Arms: Vildagliptin+metformin
Drug: Metformin only — Oral Metformin 850mg QD, up-titrated to 850mg TID is clinically indicated
  Arms: Metformin only

SUMMARY:
The purpose of this study is to demonstrate that combined vildagliptin-metformin therapy is associated with clinically significant reductions in biological markers of inflammation, pro-thrombogenicity, and atherosclerosis as compared to metformin mono-therapy in a population of diabetic patients with coronary artery disease who undergo cardiac rehabilitation.

The pre-specified established biological markers of inflammation, pro-thrombogenicity, and atherosclerosis will include: interleukin-6 (IL-6 - primary biological marker), hs-CRP, platelet reactivity testing, MMP-9, Interleukin 1 beta (IL-1 beta) and adiponectin levels.

DETAILED DESCRIPTION:
The study is designed as a single-center, randomized, non-blinded, clinical trial to provide evidence on the effects of vildagliptin on key biomarkers of atherothrombosis and inflammation. We plan to prospectively enroll 60 patients with proven coronary artery disease and randomize them in a 2:1 ratio to either vildagliptin-metformin therapy (n=40) or metformin therapy (n=20).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus on oral mono-therapy or diet only treatment
* Stable documented ischemic Heart disease (>30 days post AMI, CABG or PCI)
* Sub-optimal Hb A1c as defined ≥6.5%
* Age > 21
* Life expectancy >1 year

Exclusion Criteria:

* Significant renal impairment (creatinine ≥1.4 mg\dL females or ≥1.5 mg\dL males)
* Planned coronary intervention or planed surgical intervention (PCI or CABG)
* Planned surgical intervention
* Recent (<30 day) acute coronary syndrome (ACS)
* Hypersensitivity to either of the study drug components
* History of lactic acidosis
* Type I diabetes
* Current Hb A1c >9%
* Current Insulin treatment
* Active treatment with GLP-1 or DPP4i medication
* Hepatic impairment or ALT\AST elevations beyond X2 upper normal limit or known hepatic failure
* Inability to comply with study protocol
* Active malignancy other than basal cell carcinoma (BCC)
* Clinically advanced congestive heart failure - NYHA III-IV
* Severe left ventricular dysfunction (LVEF<30%) with NYHA II or any NYHA class with documented recent heart failure decompensation (<3 months)
* Severe stable cardiac angina CCS III - IV or Unstable angina
* Chronic inflammation (i.e. IBD, Lupus, inflammatory arthritis, rheumatoid arthritis) or chronic infection (i.e. chronic diabetic foot infection)
* Pregnancy, lactation or child-bearing potential

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reduction in serum levels of Interleukin 6 (IL-6) | 3 months

SECONDARY OUTCOMES:
Improvement in other markers of athero-thrombosis and inflammation: | 3 months
  I. Improvement in other markers of athero-thrombosis and inflammation:
  1. High sensitivity C-reactive protein (hs-CRP),
  2. Platelet reactivity
  3. Adiponectin levels
  4. IL-1 beta
  5. Matrix metallo-peptidase 9 (MMP-9)
  6. Additional exploratory markers including: IL-1 alpha ,, IL-17, TNF-alpha, MCP-1

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klempfner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Cardiac Rehabilitation Institute, Tel Litwinsky, Israel

REFERENCES:
- [Background] Shah Z, Kampfrath T, Deiuliis JA, Zhong J, Pineda C, Ying Z, Xu X, Lu B, Moffatt-Bruce S, Durairaj R, Sun Q, Mihai G, Maiseyeu A, Rajagopalan S. Long-term dipeptidyl-peptidase 4 inhibition reduces atherosclerosis and inflammation via effects on monocyte recruitment and chemotaxis. Circulation. 2011 Nov 22;124(21):2338-49. doi: 10.1161/CIRCULATIONAHA.111.041418. Epub 2011 Oct 17. PMID 22007077
- [Background] Goossen K, Graber S. Longer term safety of dipeptidyl peptidase-4 inhibitors in patients with type 2 diabetes mellitus: systematic review and meta-analysis. Diabetes Obes Metab. 2012 Dec;14(12):1061-72. doi: 10.1111/j.1463-1326.2012.01610.x. Epub 2012 May 17. PMID 22519906
- [Background] Zoungas S, Patel A, Chalmers J, de Galan BE, Li Q, Billot L, Woodward M, Ninomiya T, Neal B, MacMahon S, Grobbee DE, Kengne AP, Marre M, Heller S; ADVANCE Collaborative Group. Severe hypoglycemia and risks of vascular events and death. N Engl J Med. 2010 Oct 7;363(15):1410-8. doi: 10.1056/NEJMoa1003795. PMID 20925543
- [Background] Jenny NS, Brown ER, Detrano R, Folsom AR, Saad MF, Shea S, Szklo M, Herrington DM, Jacobs DR Jr. Associations of inflammatory markers with coronary artery calcification: results from the Multi-Ethnic Study of Atherosclerosis. Atherosclerosis. 2010 Mar;209(1):226-9. doi: 10.1016/j.atherosclerosis.2009.08.037. Epub 2009 Aug 28. PMID 19766217
- [Background] Derosa G, Maffioli P, Ferrari I, Mereu R, Ragonesi PD, Querci F, Franzetti IG, Gadaleta G, Ciccarelli L, Piccinni MN, D'Angelo A, Salvadeo SA. Effects of one year treatment of vildagliptin added to pioglitazone or glimepiride in poorly controlled type 2 diabetic patients. Horm Metab Res. 2010 Aug;42(9):663-9. doi: 10.1055/s-0030-1255036. Epub 2010 Jun 17. PMID 20560108
- [Derived] Younis A, Eskenazi D, Goldkorn R, Leor J, Naftali-Shani N, Fisman EZ, Tenenbaum A, Goldenberg I, Klempfner R. The addition of vildagliptin to metformin prevents the elevation of interleukin 1ss in patients with type 2 diabetes and coronary artery disease: a prospective, randomized, open-label study. Cardiovasc Diabetol. 2017 May 22;16(1):69. doi: 10.1186/s12933-017-0551-5. PMID 28532406